CLINICAL TRIAL: NCT04472858
Title: A Phase I, Multicenter,Open-label,Dose-Escalation and Expansion Study of CS1001 in Combination With Donafenib in Patients With Advanced Solid Tumors
Brief Title: A Study of CS1001 in Combination With Donafenib in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Collaborators: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS1001/Donafenib-101
Record Dates: First submitted 2020-07-08; First posted 2020-07-16 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cholangiocarcinoma (Experimental): Cholangiocarcinoma
  Interventions: Drug: Donafenib; Drug: CS1001
- Squamous cell carcinoma of the head and neck (Experimental): Squamous cell carcinoma of the head and neck（HNSCC）
  Interventions: Drug: Donafenib; Drug: CS1001
- Endometrial cancer (Experimental): Endometrial cancer
  Interventions: Drug: Donafenib; Drug: CS1001

INTERVENTIONS:
Drug: Donafenib — dose escalation: Donafenib 100 mg QD/100 mg BID/200 mg BID (p.o.). dose expansion: Patients will be assigned to specific tumor types and treated at the recommended dose for dose escalation.The recommended dose for dose escalation will be determined by the dose escalation study.
Drug: CS1001 — CS1001 will be administrated by intravenous (i.v.) infusion once every 28 days

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and treatment effect of CS1001 in combination with Donafenib in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This trail uses an open, multi-center study design, Contains two parts: a dose escalation part and a dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand this study and voluntarily sign ICF;
* 18 to 75 years old (including 18 and 75 years old), male or female;
* Subjects with advanced solid tumors, including:

Phase I study:

subjects with advanced solid tumors confirmed by histology or cytology that are not suitable for surgical resection, or have failed or tolerated standard treatment, or have no standard treatment. Including but not limited to Cholangiocarcinoma , head and neck squamous cell carcinoma (HNSCC) and endometrial cancer.

Exclusion Criteria:

* Any history of active autoimmune diseases or autoimmune diseases; patients with vitiligo or asthma that has been completely relieved in childhood, and patients who do not need any intervention after adulthood can be included;
* Participants with any condition that impairs their ability to take oral medication, such as lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Patients with uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage and need to retain a catheter;
* Human immunodeficiency virus (HIV) antibody positive;
* Patients who are simultaneously infected with hepatitis B virus and hepatitis C virus;
* Lactating women. If they are willing to stop breastfeeding, they can also be included in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | From the day of first dose to 21 days after last dose
To determine the dose limiting toxicity (DLT) | In the dose escalation part, from the day of first dose to 21 days after last dose
To determine the maximum tolerated dose(MTD) | In the dose escalation part, from the day of first dose to 21 days after last dose
To determine the recommended dose of phase II | In the dose escalation part, from the day of first dose to 21 days after last dose
Objective response rate as determined by the Invertigator using RECIST V1.1 | In the dose escalation part, from the day of first dose to 21 days after last dose

SECONDARY OUTCOMES:
Anti-CS1001 antibody | From the day of first dose to 21 days after last dose
Objective response rate (ORR) | From the day of first dose to 21 days after last dose
Overall survival(OS) | From the day of first dose to 21 days after last dose
Progression free survival(PFS) | From the day of first dose to 21 days after last dose
Duration of remission (DOR) | From the day of first dose to 21 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai Eastern Hospital, Shanghai, Shanghai Municipality, China